CLINICAL TRIAL: NCT06830993
Title: Development and Testing of an Innovative Patient-Centered Physical Activity Program for Hemodialysis Patients
Brief Title: Physical Activity Prescription Program for Hemodialysis Patients
Acronym: Move More
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Kenneth Wilund, Director and Professor of the School of Nutritional Science and Wellness. University of Arizona, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004405
Record Dates: First submitted 2025-02-13; First posted 2025-02-17 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Hemodialysis
Keywords: hemodialysis; physical activity; fatigue; physical function; exercise; patient reported outcome
MeSH Terms: conditions — Motor Activity; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Move More Personalized Exercise Program (Experimental): Personalized physical activity program aimed to increase the physical activity levels determined through a point system. Points are derived from metabolic equivalent (MET) scores and can be accumulated by performing any activity (e.g., "lifestyle" activities, aerobic, and/or resistance exercises) the participants complete. Weekly challenges/goals will be set to encourage participants to increase their physical activity levels. Participants will have the autonomy to decide about their weekly challenges or goals.
  Interventions: Behavioral: "Move More" Personalized Exercise Program
- Intradialytic Exercise Program (Active Comparator): Participation in an Intradialytic cycling (exercise during dialysis) physical activity prescription and resistance ("strength training") exercise for 6 months.
  Interventions: Behavioral: Intradialytic Exercise Program

INTERVENTIONS:
Behavioral: "Move More" Personalized Exercise Program — "Move More" - a personalized exercise program involving both in center and out-of-center exercise. Our novel intervention provides patient's the autonomy to choose the types of physical activity and exercise that they are willing and able to participate in. In brief, it involves working one-on-one with patients to develop an activity prescription that aims to get participants to "move more", by any means necessary.
  Arms: Move More Personalized Exercise Program
Behavioral: Intradialytic Exercise Program — Those in the intradialytic exercise group will undergo a variety of exercises including intradialytic cycling and resistance ("strength training").
  Arms: Intradialytic Exercise Program

SUMMARY:
The goal of this clinical trial is to compare the efficacy of a standard intradialytic exercise program (control group) to an individualized, patient-centered, "Move-More" physical activity intervention (intervention group) in hemodialysis (HD) patients.

Exercise programs often fail to yield robust benefits for many HD patients, in part because the type and volume of exercise prescribed is inappropriate for a variety of reasons, and the benefits from these studies are often disappointing, as they are characterized by poor adherence, high dropout rates, and modest effects on physical function, body composition, cardiovascular disease risk, and other outcomes related to quality of life (QOL). To address this, the investigators have designed a novel physical activity intervention "Move More" that is designed to overcome many of the barriers to increasing physical activity in this population. This study aims to compare the efficacy of a standard intradialytic exercise program (control group) to an individualized, patient-centered, "Move-More" physical activity intervention (intervention group) in HD patients. The investigators primary hypothesis is that patients randomized to the Move More intervention will increase their physical activity levels more than those in the intradialytic exercise group.

The main question it aims to answer is:

• Does "Move More" increase the physical activity levels (minutes) measured through weekly minutes of physical activity and the LoPAQ questionnaire more than those in the standard intradialytic exercise program?

For secondary outcomes this study aims to answer the following:

* Does "Move More" improve the physical function of hemodialysis patients assessed by the short physical performance battery (SPBB) more than those in the standard intradialytic exercise program?
* Does "Move More" decrease fatigue assess by the SONG-HD survey more than those in the standard intradialytic exercise program?
* Does "Move More" decrease symptoms of depression assessed by PROMIS Depression Short Form 8a more than those in the standard intradialytic exercise program?
* Does "Move More" increase the amount of exercise measured through a point system more than those in the standard intradialytic exercise program?
* Does "Move More" improve blood pressure (BP) more than those in the standard intradialytic exercise program?

DETAILED DESCRIPTION:
Individuals with kidney failure receiving maintenance hemodialysis (HD) have very low physical activity levels and poor physical function, and this contributes to a poor quality of life and premature mortality. To help address this problem, many researchers and clinicians have implemented simplistic physical activity programs that include mandated exercise prescriptions such as cycling during dialysis, light resistance training, or at-home walking programs. But the benefits from these studies are often disappointing, as they are characterized by poor adherence, high dropout rates, and modest effects on physical function, body composition, cardiovascular disease risk, and other outcomes related to QOL. To address this, the investigators have designed a novel physical activity intervention (Move More) that is designed to overcome many of the barriers to increasing physical activity in this population.

The goal of the program is to accumulate an increasing number of points derived from metabolic equivalent (MET) each week the participant is in the program, indicating that their physical activity levels are increasing throughout. The rationale for this approach is that participants are able to choose activities that are important to them, as opposed to prescribed mandated exercises they may not value or benefit from. In brief, it involves working one-on-one with patients to develop an activity prescription that aims to get participants to "move more", by any means necessary.

This includes developing strategies to incorporate more "lifestyle" physical activity into patients' lives (e.g., grocery shopping, yardwork, walking a dog, etc.), as well as structured exercises, including body weight exercises, flexibility training, aerobic exercise and/or recreational activities. Importantly, the activities that are prescribed are the types that they are willing and able to do. This contrasts with what is normally done, which is to assign specific types of exercise that they may not be motivated or willing to do. The investigstors recently conducted a pilot and feasibility study using this novel intervention approach in dialysis clinics in East-Central Illinois. Our preliminary results indicate that the approach is feasible to implement, and the participants were able to increase their physical activity levels to a much greater extent than is normally seen when using mandated exercise prescriptions. Qualitative data from this trial also indicated that the patients exposed to our "Move More" intervention enjoyed the program and would be willing to maintain their increased physical activity levels after the trial was over.

In this study, participants will be assessed for eligibility and following baseline testing they will be randomly assigned to one of two groups. Patients will complete a medical history form that will help assess participation eligibility. In addition, a physician clearance form must be signed by the patient's nephrologist to participate in the study. Once declared eligible for the study and cleared by their physician, patients will undergo baseline testing.

The first group (Move More) will participate solely in our personalized physical activity prescription (Move More) program. The physical activity prescription will be individualized based on the participants' needs assessment (consultation) at baseline. Exercise progression will also be made on an individual basis and be determined through a point system (METs). Points are derived from metabolic equivalent (MET) scores and can be accumulated by performing any activity (e.g., "lifestyle" activities, aerobic, and/or resistance exercises) the participants complete.

Accumulated points are based on MET values from the Physical Activity compendium. Points are derived from metabolic equivalent (MET) scores and can be accumulated by performing any activity (e.g., "lifestyle" activities, aerobic, and/or resistance exercises) the participants complete. The participants will accumulate points based on MET values from the Physical Activity compendium, which the investigators will provide. For completing 10 minutes of any activity, the participants will "earn" the number of points corresponding to that activity's published MET values. Points will be based on the actual minutes of each activity performed. For example, the published MET value for brisk walking is 3.5 METS. Based on this, the participants will receive 3.5 points for every 10 minutes of brisk walking. The overall goal is to accumulate more points each week for the duration of the intervention.

If randomized into the control group participants will undergo a variety of exercises including intradialytic cycling and resistance ("strength training") exercise. The Move More and Cycle programs will be conducted for 6 months and participants will be engaged to participate 3x/week, during participants' regularly scheduled hemodialysis treatments.

Our primary hypothesis is that patients randomized to the Move-more intervention will increase their physical activity levels more than those in the intradialytic exercise group. Physical activity levels will be assessed using weekly training logs and physical activity questionnaires at baseline and final testing (at 6 months).

At the beginning and end of the study (0 and 6 months), participants will undergo a few tests to measure their physical function, including their walking speed, their ability to rise from a chair, ("sit to stand test"), and a balance test, these tests are part of the Short Physical Performance Battery. The investigators will also provide them with a series of short questionnaires to measure their self-reported physical activity levels (LoPAQ), depression (PROMIS Depression Short Form 8a), and fatigue (SONG-HG survey). The purpose of these tests is to determine if the participants in the "Move-More" group show greater improvements in these measurements than those in the intradialytic exercise group.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old (no upper age limit);
* Chronic hemodialysis for ≥ 3 months;
* No planned or expected change in dialysis modality, elective surgery, or relocation during the study period (24 weeks);
* Able to communicate in English or Spanish and provide written informed consent;
* Assessed to be safe and able to exercise by the Hemodialysis unit nephrologist

Exclusion Criteria:

* Physical Activity: patients undergoing >150 minutes/week of prescribed PA at baseline will be excluded from the study.
* Physician Clearance: Patients who do not receive physician clearance to participate in the study will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Activity | baseline, 3 months, 6 months
  Total Minutes of Physical Activity measured with minutes, there is no a minimum or maximin value. If participants increased the total minutes of physical activity this means they increased their physical activity levels.

SECONDARY OUTCOMES:
Change in Physical Activity | baseline, 3 months, 6 months
  Low Physical Activity Questionnaire (LoPAQ). Minimum value: 0 (indicating no physical activity). Maximum value: 24 (representing the highest level of low-intensity physical activity measured by the questionnaire)
Change in Physical Activity | baseline, 3 months, 6 months
  Points derived from metabolic equivalents (METs). Points of Physical Activity measured with METs, there is not a minimum or maximin value. If participants increased their points this means they increased their physical activity levels. If they decreased their points this means they decrease their physical activity levels.
Change in Fatigue | baseline, 3 months, 6 months
  Standardized Outcomes in Nephrology - Hemodialysis Fatigue (SONG-HD Fatigue measure). Minimum Value: 0 (indicating no fatigue). Maximum Value: 10 (indicating the most severe fatigue)
Change in Depressive symptoms | baseline, 3 months, 6 months
  Patient Reported Outcomes Measurement Information System- Depression Short Form 8a (PROMIS Depression SF 8a). Minimum Value: 8 (lowest possible raw score, indicating the least depressive symptoms). Maximum Value: 40 (highest possible raw score, indicating the most severe depressive symptoms). The raw scores are typically converted into T-scores (mean = 50, SD = 10) for standardized interpretation.
Change in Physical function | baseline, 3 months, 6 months
  Short Physical Performance Battery (SPPB). Minimum Value: 0 (indicating the worst physical performance). Maximum Value: 12 (indicating the best physical performance)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth R Wilud, PhD, Principal Investigator — University of Arizona
Locations (1):
- DCI Desert Dialysis, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD used in the results publication

REFERENCES:
- [Background] Manfredini F, Mallamaci F, D'Arrigo G, Baggetta R, Bolignano D, Torino C, Lamberti N, Bertoli S, Ciurlino D, Rocca-Rey L, Barilla A, Battaglia Y, Rapana RM, Zuccala A, Bonanno G, Fatuzzo P, Rapisarda F, Rastelli S, Fabrizi F, Messa P, De Paola L, Lombardi L, Cupisti A, Fuiano G, Lucisano G, Summaria C, Felisatti M, Pozzato E, Malagoni AM, Castellino P, Aucella F, Abd ElHafeez S, Provenzano PF, Tripepi G, Catizone L, Zoccali C. Exercise in Patients on Dialysis: A Multicenter, Randomized Clinical Trial. J Am Soc Nephrol. 2017 Apr;28(4):1259-1268. doi: 10.1681/ASN.2016030378. Epub 2016 Dec 1. PMID 27909047
- [Background] Koh KP, Fassett RG, Sharman JE, Coombes JS, Williams AD. Effect of intradialytic versus home-based aerobic exercise training on physical function and vascular parameters in hemodialysis patients: a randomized pilot study. Am J Kidney Dis. 2010 Jan;55(1):88-99. doi: 10.1053/j.ajkd.2009.09.025. Epub 2009 Nov 22. PMID 19932545
- [Background] Graham-Brown MPM, March DS, Young R, Highton PJ, Young HML, Churchward DR, Dungey M, Stensel DJ, Bishop NC, Brunskill NJ, Smith AC, McCann GP, McConnachie A, Burton JO. A randomized controlled trial to investigate the effects of intra-dialytic cycling on left ventricular mass. Kidney Int. 2021 Jun;99(6):1478-1486. doi: 10.1016/j.kint.2021.02.027. Epub 2021 Apr 8. PMID 34023029
- [Background] Jeong JH, Biruete A, Tomayko EJ, Wu PT, Fitschen P, Chung HR, Ali M, McAuley E, Fernhall B, Phillips SA, Wilund KR. Results from the randomized controlled IHOPE trial suggest no effects of oral protein supplementation and exercise training on physical function in hemodialysis patients. Kidney Int. 2019 Sep;96(3):777-786. doi: 10.1016/j.kint.2019.03.018. Epub 2019 Apr 2. PMID 31200945